CLINICAL TRIAL: NCT05504967
Title: Single-center, Double-blind, Placebo-controlled Study Evaluating the Efficacy of Pre-incisional Local Analgesia With Ropivacaine and Dexamethasone for Pain Management After Tonsillectomy
Brief Title: CT Evaluating the Efficacy of Pre-incisional Local Analgesia With Ropivacaine + Dexamethasone in Pain Management After Tonsillectomy
Acronym: ORL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2CA_2019_ORL_01; 2019-000202-29 (EudraCT Number)
Record Dates: First submitted 2022-05-26; First posted 2022-08-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Tonsillectomy
Keywords: Tonsillectomy; Pain management
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dexamethasone (Active Comparator): 12.5mg dexamethasone + saline solution peramygdalin infiltration in each loca (25mg in total).
  Single dosage pre-incisional.
  Interventions: Drug: Oradexon; Drug: Saline solution
- ropivacain (Active Comparator): 18.75 mg ropivacain + saline solution peramygdalin infiltration in each loca (37mg in total).
  Single dosage pre-incisional.
  Interventions: Drug: Ropivacaine; Drug: Saline solution
- ropivacain + dexamethasone (Experimental): 18.75mg ropivacain + 12.5mg dexamethasone peramygdalin infiltration (in each loca).
  Single dosage pre-incisional.
  Interventions: Drug: Oradexon; Drug: Ropivacaine
- placebo (Placebo Comparator): Saline solution (NaCl 0.9%) peramygdalin infiltration (in each loca). Single dosage pre-incisional. 4 syringes must be prepared, two for each of the tonsil sites.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Oradexon — With a syringe aspirate 2.5 ml of a 5mg/ml dexamethasone solution, for a total of 12.5mg. Repeat the procedure with another syringe. 2 syringes must be prepared, one for each of the tonsil sites.
  Other Names: dexamethasone
  Arms: dexamethasone; ropivacain + dexamethasone
Drug: Ropivacaine — With a syringe aspirate 2.5 ml of a 7.5mg/ml dexamethasone solution, for a total of 18.75mg. Repeat the procedure with another syringe. 2 syringes must be prepared, one for each of the tonsil sites.
  Arms: ropivacain; ropivacain + dexamethasone
Drug: Saline solution — With a syringe, aspirate 2.5 ml of a 0.9% NaCl solution. Repeat the procedure with another syringe. 2 syringes must be prepared, one for each of the tonsil sites.
  Arms: dexamethasone; placebo; ropivacain

SUMMARY:
This study is a randomized, controlled, double-blind clinical trial to evaluate the effect of local infiltration of ropivacaine and dexamethasone, alone or in association, in the reduction of pain and the need for supplementary analgesia, after tonsillectomy, in the immediate and late postoperative period, in individuals aged 18 to 65 years.

The present clinical trial will include 4 study groups, each with different content of infiltration into the amygdaline locus. One group will have ropivacaine in the infiltration, the other will have dexamethasone and another the association of these two drugs. In order to better understand the effectiveness of these drugs, there will also be a control group, in which saline solution will be infiltrated.

Approximately 104 individuals, aged 18 to 65 years, proposed for tonsillectomy will be included in the study, i.e., 26 subjects in each study group.

Postoperative pain will be characterized by self-assessment through the Visual Analog Scale (VAS, 100mm) at various moments of the study, namely in the preoperative consultation, in the pre-anesthetic consultation, at hospital admission and in the postoperative period until the 15th day after the surgery.

The aim of this study is not to eliminate intra and postoperative analgesia, but rather account for the need for analgesia depending on the different infiltration content peramygdalin. For this, in the postoperative period, a careful pain monitoring, having first-line analgesic and rescue medication for use immediate response in the face of minimal pain assessed by validated pain scales. It is intended, therefore, to record which analgesic drugs and in what doses were necessary.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II;
* Surgical proposal of tonsillectomy;
* Tonsillectomy performed by the cold shedding technique;
* History of recurrent tonsillitis, caseous tonsillitis and / or peritonsillar abscess;

Exclusion Criteria:

* Use of chronic analgesic medication;
* ASA III-IV;
* Coagulation disorders, such as von Willebrand disease or diagnosis of other platelet disorders, haemophilia A and B, or diseases that may develop with hemostatic dysfunction;
* Intolerance or allergy to any of the drugs used in the study;
* Suspicious or confirmed diagnosis of neoplastic disease;
* Fever or acute respiratory tract infection in the last 3 weeks;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in pain assessment using the VAS | Change from baseline (90 days before surgery; day of surgery, day 1, 2, 3, 7 and 15 after surgery)
  Alteration in Visual Analogue Scale values (1-100mm) to assess pain at rest and during swallowing
Time to first administration of analgesia | From the day of surgery to discharge (an average 1 day)
  Time until it is needed to administer analgesia to the patient, after surgery (in minutes)
Paracetamol intake | Time since the end of surgery until post-operative visit (15 days after surgery)
  Number of paracetamol intakes
Paracetamol cumulative dosage intake | Time since the end of surgery until post-operative visit (15 days after surgery)
  Cumulative dosage of paracetamol intake in mg
Rescue analgesia intake | Time since the end of surgery until post-operative visit (15 days after surgery)
  Number of rescue analgesia intakes (tramadol)
Need of Pethidine | Immediate post-surgery
  Need of pethidine in immediate post-surgery (yes/no)
Time to need of Pethidine | Time since the end of surgery until post-operative visit (15 days after surgery)
  Time until pethidine admnistration is needed, since the end of surgery (minutes)
Time to onset of water intake, liquid and solid oral diet | Time since the end of surgery until post-operative visit (15 days after surgery)
  Time to onset of water intake, liquid and solid oral diet, since the end of surgery (minutes)

SECONDARY OUTCOMES:
Safety outcome | Time since screening until post-operative visit (15 days after surgery)
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ana Menezes, Principal Investigator — Serviço de Otorrinolaringologia, Hospital de Braga, EPE
Locations (1):
- Serviço de Otorrinolaringologia, Hospital de Braga, Braga, Portugal